CLINICAL TRIAL: NCT02397850
Title: Optimizing Psychotherapeutic Aftercare for Patients Suffering From Chronic/Recurrent Depression: Development and First Evaluation of a Telephone-based Continuation Treatment (Pilot Study).
Brief Title: Development of a Telephone-based Continuation Treatment for Patients With Chronic Depression.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WATZKE-892
Record Dates: First submitted 2015-01-14; First posted 2015-03-25 (Estimated); Last update posted 2017-11-07 (Actual); Status verified 2017-11

CONDITIONS: Chronic Depressive Disorder
Keywords: depression, chronic, psychotherapy, telephone, feasibility
MeSH Terms: conditions — Depression; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 30 min or 50 min (Experimental): Patients receive either seven 30 minutes or 50 minutes phone calls over 6 months (psychotherapy/continuation treatment)
  Interventions: Behavioral: phone calls 30 min; Behavioral: phone calls 50 min

INTERVENTIONS:
Behavioral: phone calls 30 min — Patients receive either seven 30 minutes phone calls over 6 months (psychotherapy/continuation treatment)
Behavioral: phone calls 50 min — Patients receive either seven 50 minutes phone calls over 6 months (psychotherapy/continuation treatment)

SUMMARY:
There is a high risk for relapse in people suffering from depression. Studies indicate that the continuation of an acute psychotherapeutic treatment can reduce the likelihood of relapse. Therefore, this pilot study is aimed to investigate the feasibility of a continuation psychotherapy over 6 months, to support people suffering from chronic forms of depression in their daily life. The investigated continuation therapy itself includes about one telephone call per month (therapist - patient), focussing on the integration of strategies into the patient's daily routine. The patients receive either 30 minutes or 50 minutes phone calls. On the one hand, these phone calls are supported by a workbook for patients containing psychoeducative elements, strategies and exercises. On the other hand, the therapist's work is based on a manual containing several modules and strategies. Both tools (workbook, manual) are understood as a framework, using the appropriate sections according to the patient's needs. As a result, the patients receive a continuation treatment which is appropriate and adapted to their individual situation.

The main purpose of this pilot study is to evaluate the feasibility of a telephone based psychotherapeutic continuation treatment with a small sample of 20 patients suffering from chronic depression. In case of promising results the effectiveness of this kind of treatment is going to be investigated within a comparative trial (including face-to-face intervention, no intervention).

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Diagnosis of chronic (300.4) or recurrent (296.31-3) depression (according to the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition)
* Currently in partial or full remission
* Previous psychotherapy (acute treatment; some kind of cognitive-behavioral therapy)
* adequate knowledge of German language
* in case of taking antidepressants: long-term and stable dosage (with unchanged taking since 3 months at least)

Exclusion Criteria:

* acute suicidality
* psychotic symptoms
* severe cognitive impairments
* in case of taking antidepressants: anticipated stopping medication within treatment period (6 months)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2015-02; Primary Completion 2017-05-20 (Actual); Study Completion 2017-10-25 (Actual)

PRIMARY OUTCOMES:
number of patients dropping out of treatment | 6 months
change of depressive symptoms from baseline to posttreatment | 6 months
  assessed by the Patient Health Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Birgit Watzke, Prof. Dr., Principal Investigator — University of Zurich
Locations (1):
- UniversitätsSpital Zürich Klinik für Psychiatrie und Psychotherapie Ambulatorium, Zurich, Switzerland